CLINICAL TRIAL: NCT04348214
Title: Screening and Risk Assessment of Healthcare Workers and Infection Control in University and COVID-19 Quarantine Hospitals Using Real-time Geospatial Mapping for Emergency Healthcare Resource Mobilization and Management
Brief Title: Screening & Risk Assessment of Healthcare Workers & Infection Control in University & COVID-19 Quarantine Hospitals
Acronym: SARAH
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Aya Mostafa, Associate Professor of Public health and Epidemiology, Ain Shams University
Other Study IDs: FMASU P18a/ 2020
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective investigation and screening of all HCWs working in all governmental university hospitals and the affiliated COVID-19 quarantine hospitals using an online survey and laboratory testing using rapid serological tests and PCR. To date, the Ministry of Higher Education has dedicated quarantine hospitals at the following governmental universities: Ain Shams, Cairo, Helwan, Alexandria, Mansoura, Assiut, Minia. This list may be expanded in the future. The project will be pilot tested in Ain Shams University, then extended to other universities subsequently. For risk categorization of HCWs exposed to COVID-19 virus and assessment of infection control needs, an online survey questionnaire will be administered to all HCWs in the governmental university hospitals involved in emergency and intensive care and in the provision of care for COVID-19 patients in the affiliated COVID-19 quarantine hospitals. For confirmation of infection and determination of the secondary infection rate, paired serological samples at baseline and after exposure will be collected. For measuring the validity of the available rapid serological tests, a respiratory sample will be taken for viral detection by RT-PCR. A real-time interactive map using geographical information system programming will be developed to flag hotspots for HCWs' risk and infection control needs that originated from the online survey risk categorization in governmental university and COVID-19 quarantine hospitals. Policy and decision makers will use the map to manage emergency healthcare resource mobilization based on HCWs' risk and infection control needs.

DETAILED DESCRIPTION:
Research Approach and Methodology

1. Healthcare workers' risk and 2. Infection prevention and control needs: Study design and setting

To fulfill specific objectives, a prospective investigation of all HCWs working in all governmental university hospitals and the affiliated COVID-19 quarantine hospitals.

To date, the Ministry of Higher Education has dedicated quarantine hospitals at the following governmental universities: Ain Shams, Cairo, Helwan, Alexandria, Mansoura, Assiut, Minia. This list may be expanded in the future. The project will be pilot tested in Ain Shams University, then extended to other universities subsequently.

Study population For the purpose of this study, HCWs are defined as all staff in the governmental university hospitals involved in emergency and intensive care and in the provision of care for COVID-19 patients in the affiliated COVID-19 quarantine hospitals. These include those who have been present in the same area as the patient, as well as those who may not have provided direct care to the patient, but who have had contact with the patient's body fluids, potentially contaminated items or environmental surfaces. This includes health care professionals, allied health workers, auxiliary health workers (e.g. cleaning and laundry personnel, x-ray physicians and technicians, clerks, phlebotomists, respiratory therapist, nutritionists, social workers, physical therapists, lab personnel, cleaners, admission/reception clerks, patient transporters, catering staff etc.). Once a case of COVID-19 has been identified in these hospitals, a list of all health care workers with any exposure to COVID-19 patient will need to be drawn up.

Study tool and data collection For risk categorization of HCWs exposed to COVID-19 virus and assessment of infection control needs, an online survey questionnaire will be administered to all HCWs in the governmental university hospitals involved in emergency and intensive care and in the provision of care for COVID-19 patients in the affiliated COVID-19 quarantine hospitals.

The questionnaire will be adapted from the World Health Organization relevant protocols and interim guidance. The sections of the questionnaire will cover:

1. Socio-demographic, background information including history of tobacco use, and pre-existing medical conditions;
2. COVID-19 virus exposure risk assessment for community exposure;
3. COVID-19 virus exposure risk assessment for nosocomial exposure (i.e. contact and possible exposure with the COVID-19 patients since the patient has been admitted to the health care facility);
4. HCW interactions with COVID-19 patient information;
5. HCW activities performed on COVID-19 patient in health care facility;
6. HCW symptoms;
7. Adherence to infection prevention and control measures during health care interactions;
8. Adherence to infection prevention and control measures when performing aerosol-generating procedures (e.g. tracheal intubation, nebulizer treatment, open airway suctioning, collection of sputum, tracheotomy, bronchoscopy, cardiopulmonary resuscitation, etc.); and
9. Accidents with biological material.

This online survey will be completed at baseline and at any future contact or possible exposure with the COVID-19 patients since the patient has been admitted to the hospital.

Other forms will complement the data collected in the online survey questionnaire. The complementary forms include:

* Laboratory form for specimen collection for screening and testing and the relevant results
* Follow-up laboratory form for specimen collection for screening and testing and the relevant results
* HCW symptom diary: Each HCW contact will be asked to record the presence or absence of various signs or symptoms each day for up to 21 days after the administration of the baseline questionnaire (minimum 14 days).
* Outcome form for follow up of HCWs who experience contact or possible exposure with the COVID-19 patients since the patient has been admitted to the hospital.
* Health care facility infection prevention and control form: filled once at baseline for each of the study hospitals.

These will be filled by HCWs, and dedicated teams and coordinators representing the hospital infection control focal points and the hospital management at each of the study hospitals. The forms will be electronically linked to the online survey for instant updates of HCW information using an automatically generated unique serial study number for each HCW to be used across all study forms.

3. Testing for COVID-19 among healthcare workers:

For confirmation of seroconversion, determination of the secondary-infection attack rate, and the proportion of asymptomatic infection paired serological samples will be collected:

1. A baseline serum sample will be collected from all healthcare workers with any exposure (regardless of symptoms), as soon as possible after confirmation of a COVED-19 infected patient in the hospital.
2. A second serum sample will be collected from the same healthcare workers at least 21 days after the collection of the first serum sample

For measuring the validity of the available rapid serological tests:

A respiratory sample will be taken for viral detection by RT-PCR

4. Geospatial mapping of health care workers' risk and infection control needs:

To achieve this aim the following subtasks must be done:

- Build a full stack web-based platform that is integrated with a geographical information system. Where, the platform frontend is a real-time interactive map.

Moreover, the platform backend is a database system to store and manipulate the HCWs' risk and infection control data.

* Build a real-time Signal-R flagging service to track the survey results and put flags on the platform interactive map where these flags represent the location of high HCWs' risk and infection control rate.
* Build a real-time reporting service based on Signal-R and Artificial Intelligence techniques to follow up the survey results and inform the policy and the decision makers with the location and information of the high HCWs' risk and infection control rate.

Furthermore, this reporting service provides more insights on the survey results using the Artificial Intelligence techniques such as the association between the geographical information and the high HCWs' risk rate.

ELIGIBILITY:
Inclusion Criteria:

* All staff in the governmental university hospitals involved in emergency and intensive care and in the provision of care for COVID-19 patients in the affiliated COVID-19 quarantine hospitals

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All staff in the governmental university hospitals involved in emergency and intensive care and in the provision of care for COVID-19 patients in the affiliated COVID-19 quarantine hospitals
Sampling Method: Non-Probability Sample
Enrollment: 4040 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Risk categorization of healthcare workers | 9 months
  To determine the risk categorization of HCWs for exposure to a COVID-19 patient using an online survey in governmental university and COVID-19 quarantine hospitals
COVID-19 infection rate among health care workers | 9 months
  To estimate the COVID-19 infection rate among HCWs in governmental university and quarantine hospitals.
Risk factors for COVID-19 among health care workers | 9 months
  To determine the risk factors for COVID-19 among health care workers in governmental university and quarantine hospitals.
Adherence of health care workers to infection prevention | 9 months
  To evaluate adherence of HCWs to infection prevention and control measures using an online survey in governmental university and COVID-19 quarantine hospitals.
Validity of the available rapid serological test for detecting COVID-19 virus infection | 9 months
  To determine the validity (sensitivity and specificity) of the available rapid serological test for detecting COVID-19 virus infection among HCWs in governmental university and COVID-19 quarantine hospitals.

SECONDARY OUTCOMES:
Clinical spectrum of COVID-19 | 9 months
  To characterize the risk factors, clinical spectrum, duration and severity of COVID-19 infections among HCWs in governmental university and quarantine hospitals.
Effectiveness of infection prevention in the health care facility | 9 months
  To evaluate the effectiveness of infection prevention and control measures programs at health facility level using an online survey tool in governmental university and COVID-19 quarantine hospitals
Emergency infection prevention and control needs | 9 months
  To determine the emergency infection prevention and control needs among HCWs using an online survey tool in governmental university and COVID-19 quarantine hospitals
Isolation rate and emergency health care worker replacement needs | 9 months
  To determine the isolation rate among HCWs and the need for emergency HCW replacement in governmental university and COVID-19 quarantine hospitals.
Rate of seroconversion | 9 months
  To determine the serologic response for HCWs with symptomatic and possibly asymptomatic COVID-19 virus infection in governmental university and COVID-19 quarantine hospitals.

CONTACTS AND LOCATIONS:
Overall Officials: Aya Mostafa, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mostafa A, Kandil S, El-Sayed MH, Girgis S, Hafez H, Yosef M, Saber S, Ezzelarab H, Ramadan M, Algohary E, Fahmy G, Afifi I, Hassan F, Elsayed S, Reda A, Fattuh D, Mahmoud A, Mansour A, Sabry M, Habeb P, Ebeid FS, Elanwar A, Saleh A, Mansour O, Omar A, El-Meteini M. SARS-CoV-2 seroconversion among 4040 Egyptian healthcare workers in 12 resource-limited healthcare facilities: A prospective cohort study. Int J Infect Dis. 2021 Mar;104:534-542. doi: 10.1016/j.ijid.2021.01.037. Epub 2021 Jan 20. PMID 33484863
- [Result] Mostafa A, Kandil S, El-Sayed MH, Girgis S, Hafez H, Yosef M, Saber S, Ezzelarab H, Ramadan M, Afifi I, Hassan F, Elsayed S, Reda A, Fattuh D, Mahmoud A, Mansour A, Sabry M, Habeb P, Ebeid FS, Saleh A, Mansour O, Omar A, El-Meteini M. Universal COVID-19 screening of 4040 health care workers in a resource-limited setting: an Egyptian pilot model in a university with 12 public hospitals and medical centers. Int J Epidemiol. 2021 Mar 3;50(1):50-61. doi: 10.1093/ije/dyaa173. PMID 33094320